CLINICAL TRIAL: NCT00410215
Title: A Randomized Controlled Trial Comparing Picosalax and Oral Sodium Phosphate for Colon Cleansing Prior to Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Lawrence Hookey, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hookey picosalax
Record Dates: First submitted 2006-12-08; First posted 2006-12-12 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Bisacodyl; sodium phosphate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): sodium phosphate
  Interventions: Drug: sodium phosphate
- 2 (Active Comparator): picosalax
  Interventions: Drug: picosalax
- 3 (Active Comparator): picosalax plus bisacodyl
  Interventions: Drug: picosalax plus bisacodyl

INTERVENTIONS:
Drug: picosalax plus bisacodyl — 10 mg bisacodyl three and two nights prior to colonoscopy, followed by two sachets picosalax
  Arms: 3
Drug: picosalax — two sachets of picosalax taken orally the day prior to colonoscopy
  Arms: 2
Drug: sodium phosphate — two 45 ml bottles of sodium phosphate the day prior to colonoscopy
  Arms: 1

SUMMARY:
Colon cleansing prior to colonoscopy is critically important to ensure effective colonoscopy for colon cancer screening, which is now widespread in North America. Currently available colon cleansing agents are limited either by potential safety concerns or significant limitations in the ability of patients to tolerate the preparation. Pico-salax has recently been introduced in Canada as an alternative agent and is being used more and more widely despite an almost complete lack of clinical data supporting efficacy and safety. This study will establish the relative efficacy and patient tolerability of this agent and its safety profile. This is a very important, practical issue which continues to challenge gastroenterologists, surgeons, internists, family doctors and thousands of their patients in Canada on a daily basis.

Anecdotal evidence suggests that the efficacy of pico-salax when used as a sole agent may not be as efficacious as oral sodium phosphate. Hence, our hypothesis is that the combination of pico-salax and bisacodyl will provide the most efficacious bowel preparation in comparison with oral sodium phosphate and pico-salax alone, while being equally if not better tolerated.

DETAILED DESCRIPTION:
This is a randomized, investigator blinded clinical trial assessing the cleansing efficacy (using the Ottawa Bowel Preparation scale) and tolerance of three bowel cleansing regimens, two of which involve pico-salax.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive male and non-pregnant female patients
* ≥ 18 years old
* who require outpatient colonoscopy will be approached to consider participation in the study.

Exclusion Criteria:

* ileus or bowel obstruction;
* previous colorectal surgery;
* renal impairment;
* pregnancy;
* recent (<6 months) myocardial infarction or unstable angina.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2006-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Ottawa Bowel Preparation scale | At Colonoscopy.

SECONDARY OUTCOMES:
Tolerance-Likert scale questionnaire | After Preparation.
Safety Hemodynamics, Blood Chemistry | After Preparation.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence C Hookey, MD, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada